CLINICAL TRIAL: NCT05161468
Title: Bayesian Non-inferiority Trial of Injection Therapies for Acromioclavicular Joint Pain: a Randomized Clinical Trial
Brief Title: Platelet-rich Plasma, Corticosteroid, or Lidocaine for Acromioclavicular Joint Pain
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding limitation did not allow the trial to run to completion
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: The Geneva Foundation (Other); Uniformed Services University of the Health Sciences (U.S. Federal Agency); Madigan Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dan Rhon, Director, Primary Care Musculoskeletal Research Program, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 221073
Record Dates: First submitted 2021-11-19; First posted 2021-12-17 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Acromioclavicular Sprain
Keywords: acromioclavicular joint; shoulder pain; platelet rich plasma; corticosteroid
MeSH Terms: conditions — Shoulder Pain | interventions — Lidocaine; Adrenal Cortex Hormones; Triamcinolone Acetonide; Glucocorticoids; Injections; acid citrate dextrose

STUDY DESIGN:
Intervention Model Description: Bayesian regression model
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lidocaine (Active Comparator): 50 Subjects will be randomized to this group and will receive a lidocaine injection in their ACJ.
  Interventions: Drug: Lidocaine injection
- Corticosteroid (Active Comparator): 50 Subjects will be randomized to this group and will receive a corticosteroid injection in their ACJ.
  Interventions: Drug: Corticosteroid Injection
- Platelet Rich Plasma (PRP) (Active Comparator): 50 Subjects will be randomized to this group and will receive a PRP injection in their ACJ.
  Interventions: Drug: Protein Rich Plasma(PRP) Injection

INTERVENTIONS:
Drug: Lidocaine injection — 2ml of 1% lidocaine will be drawn into a 3 ml syringe and labeled. It will then be delivered into the AC joint per standard injection procedures (estimated 1-2 ml).
  Other Names: xylocaine
  Arms: Lidocaine
Drug: Corticosteroid Injection — 1 ml of triamcinolone acetonide (40 mg/ml) will be drawn with 1 ml normal saline into a 3 ml syringe and labeled. It will then be delivered into the AC joint per standard injection procedures (estimated 1-2 ml).
  Other Names: triamcinolone acetonide; glucocorticoid
  Arms: Corticosteroid
Drug: Protein Rich Plasma(PRP) Injection — 30 ml of acid-citrate-dextrose (ACD) will be drawn into a 30 ml syringe to coat the syringe. 3 ml will be left in the syringe and then 27 ml of blood will be drawn via standard venipuncture. The 30 ml mixture of blood and ACD will then be prepared in the Peak PRP system as described in the manufacturer's instruction (PEAK® PRP System). After preparation, PRP will be withdrawn (2 mls) into a 3 ml syringe and labeled. It will then be delivered into the AC joint per standard injection procedures (estimated 1-2 ml).
  Other Names: acid-citrate-dextrose (ACD)
  Arms: Platelet Rich Plasma (PRP)

SUMMARY:
This study will compare three different treatment injections for the management of acromioclavicular joint dysfunction (ACJ Dysfunction). Patients that consent and enroll will be randomized to receive (1) a corticosteroid injection, (2) an injection of Platelet Rich Plasma, or (3) a Lidocaine injection. Follow-up will occur over a 1 year period.

DETAILED DESCRIPTION:
Subjects with a diagnosis of AC joint dysfunction will be recruited through the primary care and orthopaedic clinics at participating hospitals and clinics. Patients that consent and enroll will be randomized to receive (1) a corticosteroid injection, (2) an injection of Platelet Rich Plasma, or (3) a Lidocaine injection. The primary outcome will be the change in PROMIS Physical Function Scale at 6 months post-enrollment. Secondary outcomes will include additional time points (viz, 1, 2, 3, 4, 5, and 12 months post-enrollment) and additional metrics (eg, AUC) as well as the PROMIS Pain Interference, Patient Acceptable Symptom State, Global Rating of Change, total limited duty days, and perceived recovery. Since the sample size is too small to establish non-inferiority by traditional hypothesis testing, a fully Bayesian approach will be used.

ELIGIBILITY:
Inclusion Criteria:

* TRICARE eligible beneficiaries (active duty, dependents, and military retired) with a primary complaint of AC joint pain.
* Age 18-65 years
* Able to speak and read English well enough to provide informed consent, follow study instructions and independently answer the questionnaires/surveys.
* Tender to palpation over the AC joint that reproduces the specific pain they are seeking care for
* Provocative test (cross-arm test, pain with push-ups, etc) that reproduces the specific pain they are here to seek care for

Exclusion Criteria:

* In the last year, the subject received any invasive interventions including injections (corticosteroid, hyaluronic acid, lidocaine, PRP, etc.) or surgery for the affected shoulder - specifically to the AC joint.
* Anyone separating from the military within 10 months (other than normal military retirement), pending a medical evaluation board, discharge from the military for medical reasons, or pending or undergoing any litigation for an injury
* AC Joint separation that are with a severity of Grades III-VI (in most cases, these are treated surgically, although 78% of military surgeons recommended preferring conservative care for Grade III separations, and 86% recommending at least 3 months of conservative care before surgical consideration.
* Systemic Disease that could otherwise be responsible for the shoulder pain (i.e. rheumatoid arthritis, gout, or psoriatic arthritis), non-musculoskeletal conditions causing shoulder pain, personal history of neoplasm, current or recent shoulder joint infection, acute fracture or dislocation of the shoulder related to the current episode of pain, or other more likely primary musculoskeletal shoulder disorders (rotator cuff pathology, bicipital tendonitis, etc.)
* Concurrent adhesive capsulitis of the affected shoulder
* History of intolerance or allergy to corticosteroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Patient Reported Outcomes Measurement Information Systems (PROMIS) - Physical Function Scale Computer Adapted Test (PF-CAT) | 6 months
  The PROMIS PF-CAT uses a 121-item bank to assess current self-reported capabilities related to physical activities. Like all PROMIS measures, the measure is reported on a T score metric, with a score of 50 aligning with the general population mean and a standard deviation of 10. Higher scores indicate more of the quantity being assessed.

SECONDARY OUTCOMES:
Patient Acceptable Symptom Scale (PASS) | 6 months
  We will use the PASS as a global, dichotomized single-item score indicating if patients are satisfied with the current state of their symptoms. This tool has been validated in patients with osteoarthritis. The PASS asks the patient; "Taking into account all the activities you have during your daily life, your level of pain, and also your functional impairment, do you consider that your current state is satisfactory?" Response options are "yes" or "no"
Global Rating of Change (GROC) | 6 months
  The GROC measures changes in perceived quality of life, in a variety of pain populations. It has a 15-point scale (-7 to +7), with a 0 indicating 'about the same", a -7 indicating 'a very great deal worse', and a +7 indicating a 'a very great deal better'. A score of -2 (a little bit worse) to +2 (a little bit better) indicates a perception of no change in the condition from baseline. A+3 ('somewhat better') or higher demonstrates a clinically significant improvement.
EuroQoL (EQ-5D) | Baseline; 6 Months and 1 Year after Enrollment
  the EQ-5D is a generic quality of life questionnaire that will assess quality of life on a scale that can be referenced to other disease conditions. The EQ-5D covers 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain has 3 response categories: level 1, "no problems"; level 2, "some problems"; and level 3, "inability or extreme problems." Responses are combined to give a 5-digit descriptive health state classification (e.g., 11222) The EQ-5D yields a total of 243 possible health states. Valuations for each health state are available. The EQ-5D is commonly used in economic evaluation of interventions and cost-effectiveness analysis.
Shoulder Related Costs | The 1 Year Period After Enrollment
  We will use the Military Data Repository (MDR) to identify shoulder-related healthcare costs over the 1-year follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rhon, DSc, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (2):
- United States (2):
  - Brooke Army Medical Center, San Antonio, Texas
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No
De-identified research data will be shared with Military Injury Rehabilitation Research for Operational Readiness (MIRROR) and maintained indefinitely for possible use in future research.

REFERENCES:
- [Background] Pallis M, Cameron KL, Svoboda SJ, Owens BD. Epidemiology of acromioclavicular joint injury in young athletes. Am J Sports Med. 2012 Sep;40(9):2072-7. doi: 10.1177/0363546512450162. Epub 2012 Jun 15. PMID 22707749
- [Background] Petron DJ, Hanson RW Jr. Acromioclavicular joint disorders. Curr Sports Med Rep. 2007 Oct;6(5):300-6. PMID 17883965
- [Background] Park KD, Kim TK, Lee J, Lee WY, Ahn JK, Park Y. Palpation Versus Ultrasound-Guided Acromioclavicular Joint Intra-articular Corticosteroid Injections: A Retrospective Comparative Clinical Study. Pain Physician. 2015 Jul-Aug;18(4):333-41. PMID 26218936
- [Background] Krill MK, Rosas S, Kwon K, Dakkak A, Nwachukwu BU, McCormick F. A concise evidence-based physical examination for diagnosis of acromioclavicular joint pathology: a systematic review. Phys Sportsmed. 2018 Feb;46(1):98-104. doi: 10.1080/00913847.2018.1413920. Epub 2017 Dec 13. PMID 29210329
- [Background] Wu PI, Diaz R, Borg-Stein J. Platelet-Rich Plasma. Phys Med Rehabil Clin N Am. 2016 Nov;27(4):825-853. doi: 10.1016/j.pmr.2016.06.002. PMID 27788903
- [Background] Schneider A, Burr R, Garbis N, Salazar D. Platelet-rich plasma and the shoulder: clinical indications and outcomes. Curr Rev Musculoskelet Med. 2018 Dec;11(4):593-597. doi: 10.1007/s12178-018-9517-9. PMID 30196385
- [Background] Chahla J, Cinque ME, Piuzzi NS, Mannava S, Geeslin AG, Murray IR, Dornan GJ, Muschler GF, LaPrade RF. A Call for Standardization in Platelet-Rich Plasma Preparation Protocols and Composition Reporting: A Systematic Review of the Clinical Orthopaedic Literature. J Bone Joint Surg Am. 2017 Oct 18;99(20):1769-1779. doi: 10.2106/JBJS.16.01374. PMID 29040132
- [Background] Nguyen RT, Borg-Stein J, McInnis K. Applications of platelet-rich plasma in musculoskeletal and sports medicine: an evidence-based approach. PM R. 2011 Mar;3(3):226-50. doi: 10.1016/j.pmrj.2010.11.007. PMID 21402369

DOCUMENTS (1):
  • Informed Consent Form (2022-08-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT05161468/ICF_001.pdf